CLINICAL TRIAL: NCT04227886
Title: A Prospective, Observational, Multicenter Study on Biomarkers for Predicting the Efficacy and Toxicities of Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer Based on Tissue and Plasma Exosome RNA
Brief Title: Study on Predictive Biomarkers of Neoadjuvant Chemoradiotherapy for Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhu Ji, Clinical Professor, Fudan University
Other Study IDs: FDRT-011
Record Dates: First submitted 2019-12-30; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Rectal Neoplasm Malignant Carcinoma; Chemoradiotherapy; Neoadjuvant Therapy; Predictive Biomarkers; Adenocarcinoma
Keywords: Neoadjuvant Chemoradiation; Prediction Model; Treatment Response; Toxicities; Irinotecan; Tissue RNA; Plasma exosome
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma | interventions — Radiation; capecitabine-irinotecan combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy samples and peripheral blood samples are collected before neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Good response: TRG of 0-1 is defined as good response.
  Interventions: Radiation: Radiation; Drug: Capecitabine-Irinotecan Combination
- Poor response: TRG of 2-3 is defined as poor response.
  Interventions: Radiation: Radiation; Drug: Capecitabine-Irinotecan Combination
- Light toxicity: No grade 3-4 toxicities occur during neoadjuvant therapy.
  Interventions: Radiation: Radiation; Drug: Capecitabine-Irinotecan Combination
- Heavy toxicity: Grade 3-4 toxicities occur during neoadjuvant therapy.
  Interventions: Radiation: Radiation; Drug: Capecitabine-Irinotecan Combination

INTERVENTIONS:
Radiation: Radiation — Neoadjuvant radiotherapy consisted of 50 Gy in 25 fractions using intensity-modulated radiotherapy to the primary tumor and to mesorectal, presacral, and internal iliac lymph nodes.
Drug: Capecitabine-Irinotecan Combination — The concurrent chemotherapy consists of capecitabine 625 mg/m2 twice daily 5 days per week and combined with weekly irinotecan. The irinotecan dose was used based on UGT1A1 genotype of 80mg/m2 for UGT1A1*1*1 or 65mg/m2 for UGT1A1*1*28 weekly, followed by a cycle of XELIRI.

SUMMARY:
Backgrounds: A multicenter randomized phase III trial (NCT02605265) proved that adding irinotecan guided by UGT1A1 to capecitabine-based neoadjuvant chemoradiotherapy significantly increases complete tumor response. The treatment toxicities were increased but tolerable.

Purposes: This study aims to identify the predictive biomarkers (from patients' tumor biopsy samples and peripheral blood samples before neoadjuvant therapy) for predicting the response and toxicities to neoadjuvant therapy to stratify patients and optimize treatment strategy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* Establish a predictive model for response based on tissue RNA and plasma exosome RNA
* Establish a predictive model for toxicities based on tissue RNA and plasma exosome RNA

Secondary:

* Internal validation of the established predictive models
* External validation of the established predictive models

OUTLINE:

-Treatment: Patients receive neoadjuvant therapy and surgery per the protocol. Samples collection Tumor tissue and peripheral blood will be collected prior to neoadjuvant therapy.

-Grouping: Response: Patients will be dichotomized into two groups based on the TRG. TRG of 0-1 is defined as good response. TRG of 2-3 is defined as poor response.

Toxicities: Patients will be dichotomized into two groups based on the grade of AEs. No grade 3-4 toxicities occurs during neoadjuvant therapy is defined as light toxicities. Grade 3-4 toxicities occur during neoadjuvant therapy is defined as heavy toxicities.

-Predictive Model Construction: Using RNA sequencing method to obtain the whole genome transcription profiles of the tumor tissue and plasm exosome RNA. Compare the gene expression differences between the two response groups and the two toxicity groups. Predictive models of response and toxicities are constructed.

-Internal Validation: Patients treated at Fudan University Shanghai Cancer Center (N=50) per the protocol will be enrolled as the internal validation cohort. Samples of tissue and plasm will be collected and analyzed. The performance of the model will be evaluated by the correlation of the predicted response/toxicities and the actual response/toxicities.

-External Validation: Patients treated at Liao'ning Cancer Hospital & Institute (N=50) and Harbin Medical University Cancer Hospital (N=50) per the protocol will be enrolled as two external validation cohorts. Samples of tissue and plasm will be collected and analyzed. The performance of the model will be evaluated by the correlation of the predicted response/toxicities and the actual response/toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed adenocarcinoma
* Clinical stage T3-4 andor N+
* The distance from anal verge less than 12 cm
* No suspicious metastatic disease (M1)
* ECOG PS 0-1
* UGT1A1*28 6/6 or 6/7
* No previous anti-cancer therapy

Exclusion Criteria:

* Pregnancy or breast-feeding women
* Serious medical illness
* Baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage T3 or T4 and/or N+ rectal adenocarcinoma cancer eligible for neoadjuvant chemoradiation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
TRG | Surgery scheduled 6-8 weeks after the end of neoadjuvant therapy
  Tumor regression grade
Toxicities | Up to 2 years
  Number of participants with chemoradiation-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Overall Survival | 3 years
  The total survival time of the participants from joining the group to the death
Progression-free Survival | 3 years
  The time period that from participants joining the groups to the progression of disease (recurrence or metastasis) or death of any cause.
Local Control rate | 3 years
  The time period that from participants joining the groups to the date of first documented pelvic failure.
pCR | Surgery scheduled 6-8 weeks after the end of neoadjuvant therapy
  Pathologic Complete Response

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No